CLINICAL TRIAL: NCT00390611
Title: A Randomized Phase II Study of Paclitaxel/Carboplatin With or Without Sorafenib in the First-Line Treatment of Patients With Stage III/IV Epithelial Ovarian Cancer
Brief Title: Paclitaxel and Carboplatin With Or Without Sorafenib In The First-Line Treatment Of Patients With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GYN 19; SR05-918
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Sorafenib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel/Carboplatin/Sorafenib (Active Comparator): Paclitaxel 175 mg/m2 1-3 hour IV infusion, Day 1 Carboplatin AUC 6 infused over 20 minutes IV, Day 1 Sorafenib 400mg PO bid
  Interventions: Drug: Sorafenib; Drug: Paclitaxel; Drug: Carboplatin
- Paclitaxel/carboplatin (Active Comparator): Paclitaxel 175 mg/m2 1-3 hour IV infusion, Day 1 Carboplatin AUC 6 infused over 20 minutes IV
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Sorafenib
  Other Names: BAY 43-9006
  Arms: Paclitaxel/Carboplatin/Sorafenib
Drug: Paclitaxel — Paclitaxel
Drug: Carboplatin — Carboplatin

SUMMARY:
This trial will compare the efficacy and toxicity of standard first-line chemotherapy alone vs. standard chemotherapy plus sorafenib in patients with stage III/IV ovarian cancer following cytoreductive surgery. Patients with residual large volume disease and/or bowel involvement will be excluded, to minimize the risk of bowel perforation.

DETAILED DESCRIPTION:
All patients must be at least 4 weeks from cytoreductive surgery before starting treatment. Patients will be randomized to receive treatment with either paclitaxel/carboplatin + sorafenib or paclitaxel/carboplatin. Paclitaxel/carboplatin will be repeated every 21 days for a maximum of 6 cycles. Patients with objective response/stable disease after completing 6 courses of chemotherapy will continue sorafenib until disease progression or for a total of 12 months.

- Regimen A:

Paclitaxel 175 mg/m2 1-3 hour IV infusion, Day 1

Carboplatin AUC 6 infused over 20 minutes IV, Day 1

Sorafenib 400mg PO bid

- Regimen B:

Paclitaxel 175mg/m2, 1-3 hour IV infusion, Day 1

Carboplatin AUC 6.0, 20 minute IV infusion, Day 1

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, stage III or IV epithelial ovarian carcinoma
2. No previous treatment with chemotherapy or radiation therapy
3. All patients must have undergone cytoreductive surgery, with the

   following results:
   1. No residual tumor nodule > 3cm
   2. No residual tumor involvement of the bowel (ie. invasion into bowel

      wall)
   3. No residual intestinal obstruction
4. Measurable or evaluable disease. Patients with elevated CA-125 levels

   and/or evaluable disease per RECIST criteria are eligible.
5. ECOG performance status 0 or 1.
6. ANC ≥ 1500/µL, platelets ≥ 100,000/µL, hemoglobin ≥ 9.0 g/dL.
7. Total bilirubin ≤ 1.5 x upper limits of normal (ULN), ALT and AST ≤ 2.5 x

   ULN (≤ 5 x ULN for patients with liver metastases)
8. Serum creatinine _ 1.5 x ULN
9. INR < 1.5 or a PT/PTT within normal limits. Patients receiving anticoagulation

   treatment with an agent such as warfarin or heparin may be

   allowed to participate. For patients on warfarin, the INR may be > 1.5,

   and should be measured prior to initiation of sorafenib and monitored at

   least weekly until INR is stable in the desired therapeutic range.
10. Women of childbearing potential must have a negative serum pregnancy

    test performed within 7 days prior to start of treatment.
11. Patients must be able to understand the nature of this study and give

written informed consent.

Exclusion Criteria:

1. Age < 18 years
2. Active cardiac disease, including: A) congestive heart failure > class II

   NYHA , B) unstable angina or onset of angina within last 3 months, C) myocardial infarction within 6 months
3. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
4. Patients with CNS metastases. Patients with neurological symptoms

   must undergo a CT scan/MRI of the brain to exclude brain metastasis.
5. Uncontrolled hypertension defined as systolic blood pressure > 150mmHg or diastolic pressure > 90mmHg, despite optimal medical management
6. Known HIV, chronic hepatitis B or chronic hepatitis C infections
7. Women who are pregnant or lactating. Women of childbearing potential

   must agree to use adequate contraception from time of study entry until

   at least 3 months after the last administration of study drug.
8. Active clinically serious infection (> grade 2)
9. Thrombotic or embolic events such as cerebral vascular accident

   including transient ischemic attacks within the last 6 months.
10. Pulmonary hemorrhage/bleeding event ≥ grade 2 within 4 weeks of

    starting treatment.
11. Any other hemorrhage/bleeding event ≥ grade 3 within 4 weeks of

    starting treatment
12. Serious non-healing wound, ulcer, or bone fracture
13. Evidence of history of bleeding diathesis or coagulopathy
14. Major surgery, open biopsy, or significant traumatic injury within 4 weeks

    of starting treatment.
15. Any condition that impairs the ability to swallow whole pills
16. Patients with any type of malabsorption
17. Known or suspected allergy to any of the agents used in this treatment
18. Use of St. John's Wort or rifampin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-10; Primary Completion 2012-07 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (17):
- United States (17):
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Medical College of Georgia Cancer Specialists, Augusta, Georgia
  - Providence Medical Group, Terre Haute, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Oncology Hematology Care, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Tennessee Valley Clinical Research, Chattanooga, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Center, Newport News, Virginia

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Period: 6 Cycles of Study Treatment
Arm/Group | Paclitaxel/Carboplatin/Sorafenib | Paclitaxel/Carboplatin
Started | 43 | 42
Completed | 34 | 37
Not Completed | 9 | 5
Period: Maintenance Sorafenib to Month 12
Arm/Group | Paclitaxel/Carboplatin/Sorafenib | Paclitaxel/Carboplatin
Started | 23 (11 patients came off-study between the end of cycle 6 and the start of maintenance) | 0 (Patients in the Paclitaxel/carboplatin arm did not recieve maintenance sorafenib)
Completed | 13 | 0
Not Completed | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Paclitaxel/Carboplatin/Sorafenib: Paclitaxel 175 mg/m2 1-3 hour IV infusion, Day 1 Carboplatin AUC 6 infused over 20 minutes IV, Day 1 Sorafenib 400mg PO bid
  Sorafenib
  Paclitaxel: Paclitaxel
  Carboplatin: Carboplatin
- Total: Total of all reporting groups
Arm/Group | Paclitaxel/Carboplatin/Sorafenib | Paclitaxel/Carboplatin | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Median (Full Range); unit: years] | 63 [31 to 78] | 62 [42 to 80] | 62 [31 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 85
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 42 | 85

OUTCOME MEASURES:

1. Primary Outcome: 2-year Progression-free Survival
Description: The proportion of patients with progression-free survival at 2 years. Progression-free survival is measured from Day 1 of study drug administration to disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death on study. Progression is defined in RECIST v1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel/Carboplatin/Sorafenib | Paclitaxel/Carboplatin
Number analyzed (Participants) | 43 | 42
percentage of participants | 40 | 40

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Number of patients with either complete response (CR) or partial response (PR) as defined in Response Evaluation Criteria in Solid Tumors (for patients with measurable disease) or determined by CA-125 levels (for patients without measurable disease). Complete Response: Disappearance of all target lesions, disappearance of all non-target lesions, and normalization of CA-125 for at least 4 weeks. In patients who have only elevated CA-125, the CA-125 must normalize (< 23U/mL) for more than 4 weeks. Partial Response: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameters. For patients with elevated CA-125 only, partial response will be defined as a > 50% decrease in the serum CA-125 level.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Paclitaxel/Carboplatin/Sorafenib | Paclitaxel/Carboplatin
Number analyzed (Participants) | 43 | 42
participants | 29 | 31

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was measured from the date of study entry until the date of death
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel/Carboplatin/Sorafenib | Paclitaxel/Carboplatin
Number analyzed (Participants) | 43 | 42
months | 36.5 [30.9 to 43.0] | NA [29.7 to NA] — Median OS and upper bound of 95% confidence interval not reached for this arm

4. Secondary Outcome: Toxicity of Paclitaxel/Carboplatin vs. Paclitaxel/Carboplatin/Sorafenib
Description: Number of patients experiencing treatment-related adverse events
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Paclitaxel/Carboplatin/Sorafenib | Paclitaxel/Carboplatin
Number analyzed (Participants) | 43 | 42
participants
  Neutropenia | 28 | 33
  Anemia | 29 | 30
  Thrombocytopenia | 26 | 25
  Febrile neutropenia | 3 | 1
  Nausea/vomiting | 33 | 37
  Peripheral neuropathy | 31 | 28
  Fatigue | 29 | 32
  Skin rash | 41 | 3
  Diarrhea | 22 | 8
  Pain-muscle | 12 | 14
  Hypersensitivity reaction (paclitaxel) | 6 | 1
  Mucositis | 16 | 7
  Constipation | 7 | 14
  Pain-joint | 9 | 11
  Anorexia | 9 | 8
  Hand-foot syndrome | 16 | 0
  Abdominal pain | 9 | 5
  Weakness | 7 | 6
  Hypertension | 10 | 2
  Dizziness | 6 | 6
  Fever (no neutropenia) | 6 | 5
  Dehydration | 5 | 4
  Dyspnea | 3 | 5
  Headache | 5 | 3
  Edema | 3 | 2
  Hyponatremia | 4 | 0
  Pruritus | 3 | 1

ADVERSE EVENTS:
Arm/Group | Paclitaxel/Carboplatin/Sorafenib | Paclitaxel/Carboplatin
Serious Adverse Events (participants affected / at risk) | 12/43 | 10/42
Other Adverse Events (participants affected / at risk) | 43/43 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel/Carboplatin/Sorafenib (N=43) | Paclitaxel/Carboplatin (N=42)
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Allergic reaction (Immune system disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Gastrointestinal disorders - Other, small bowel obstruction (Gastrointestinal disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Gastrointestinal disorders - Other, hemorrhage (Gastrointestinal disorders) | 0 | 1
General disorders and administration site conditions - Other, disease progression (General disorders) | 1 | 0
General disorders and administration site conditions - Other, failure to thrive (General disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Infusion related reaction (General disorders) | 1 | 0
Investigations - Other, pancytopenia (Investigations) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Metabolism and nutrition disorders - Other, electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel/Carboplatin/Sorafenib (N=43) | Paclitaxel/Carboplatin (N=42)
Gastrointestinal disorders - Other, nausea/vomiting (Gastrointestinal disorders) | 32 | 35
Fatigue (General disorders) | 27 | 33
Anemia (Blood and lymphatic system disorders) | 27 | 29
Peripheral sensory neuropathy (Nervous system disorders) | 28 | 28
Platelet count decreased (Blood and lymphatic system disorders) | 26 | 25
White blood cell decreased (Blood and lymphatic system disorders) | 22 | 25
Neutrophil count decreased (Blood and lymphatic system disorders) | 19 | 20
Rash (Skin and subcutaneous tissue disorders) | 35 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 21
Diarrhea (Gastrointestinal disorders) | 21 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 14
Constipation (Gastrointestinal disorders) | 7 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 11
Anorexia (Metabolism and nutrition disorders) | 9 | 9
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 8
Dizziness (Nervous system disorders) | 1 | 12
Hypertension (Vascular disorders) | 10 | 2
Fever (General disorders) | 5 | 6
Headache (Nervous system disorders) | 6 | 3
Mucositis (Gastrointestinal disorders) | 6 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Allergic reaction (Immune system disorders) | 7 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Dysgeusia (Nervous system disorders) | 3 | 4
Gastrointestinal disorders - Other, mouth ulcer (Gastrointestinal disorders) | 2 | 4
Edema (General disorders) | 3 | 2
Oral pain (Gastrointestinal disorders) | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Gastrointestinal disorders - Other, stomatitis (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites